CLINICAL TRIAL: NCT02488161
Title: Risk Factors of Adverse Outcomes at Short and Medium Term, and Development of Predictive Models, in Patients With Colorectal Cancer. IRYSS-coordinated Multicenter Study
Brief Title: Factors Related to Adverse Events in Colorectal Cancer
Acronym: CARESS-CCR
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Fondo de Investigacion Sanitaria (Other); Departamento de Sanidad del Gobierno Vasco (País Vasco, Spain) (Unknown)
Responsible Party: Principal Investigator, JOSE M QUINTANA-LOPEZ, MD PhD, PhD, Hospital Galdakao-Usansolo
Other Study IDs: PS09/00314; PS09/00910 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PS09/00746 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PS09/00805 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PI09/90460 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PI09/90490 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PI09/90453 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PI09/90441 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PI09/90397 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); 2010111098 (Other Grant/Funding Number: Departamento de Sanidad del Gobierno Vasco (País Vasco, Spain)); PI13/01692 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain)); PI13/00013 (Other Grant/Funding Number: Fondo de Investigación Sanitaria (Madrid, Spain))
Record Dates: First submitted 2015-06-16; First posted 2015-07-02 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Risk factors; Adverse events; Predictive models
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Fragments of colon or rectum obtained in the surgical intervention
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with colorectal cancer: One cohort of patients with colorectal cancer, studied before the intervention, and one month, one year, two years, three years and five years after.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Coordinated multi-center project with several complementary goals in each one of the sub-projects included. Objectives: 1.To determine risk factors of death, or major complications in the short term; 2.To determine risk factors of death, tumor recurrence, major complications, readmission or deterioration of quality of life in the mid term; 3.Evaluation of patient reported outcomes from before the intervention to the end of the follow-up. 4.To study the role of immunohisto-chemistry markers in the prediction of similar adverse results. This sub-project (coordinator) will approach the determination of risk factors of death, tumor recurrence, major complications, readmission and deterioration of quality of medium term life (1-2 years). Methodology. Design: prospective cohort study with 2 years follow-up after the surgical intervention. Participant centers: 18 hospitals of 6 Autonomous Communities of all Spain. Patients diagnosed of colorectal cancer surgically intervened. Variables: pre-intervention, those of the hospital admission, sociodemographic, immunohisto-chemistry and clinical parameters, that could be in relation to the outcomes to study. Statistic analysis: a derivation sample will be created where the possible predicting parameters will be identified, by cancer of colon or rectum. Predictive models will be created with a good discriminative capacity. A validation of those models will be performed in a validation sub-sample. Logistic and Cox regression models will be used. Simulation models for the prediction of discreet events in the long term will be used.

DETAILED DESCRIPTION:
This prospective cohort study included patients drawn from 22 hospitals belonging to the Spanish National Health Service (SNS), which covers the majority (99.8%) of the population of Spain. All covered residents have free access to their primary care physician and to the emergency departments of the hospitals. All of the hospitals have similar technological and human resources.

Patients with a diagnosis of colon cancer attending the surgical services of any of these hospitals to undergo surgery between June 2010 and December 2012 were informed of the goals of the study and invited to voluntarily participate. In order to take part in the study, a patient had to provide informed consent. All information was kept confidential. The Institutional Review Boards of the participating hospitals approved this project.

Data collected Data collected upon hospital admission included information on sociodemographic data, clinical data (including information about onset of symptoms, habits, personal and family background, comorbidities, diagnostic tests, pre-intervention treatments), preoperative data (including analytical, tumor markers and diagnostic tests), data of the outpatient anesthesia data on the surgical intervention, pathology data, and data related to the remaining days of admission (including the presence of complications, need for reintervention or death). Subsequently, data were collected up to 30 days after surgery (analytical, diagnostic tests, presence of complications, readmissions, reintervention or death). Finally, information was collected through the year including need for radiation therapy, chemotherapy (treatment schedule, cycles, complications of treatment, supportive care), laboratory results and diagnostic tests performed, presence of complications, tumor recurrence, readmission or reintervention and death.

Patients completed the following questionnaires before surgery and one year after surgery: EuroQol-5D, EORTC QLQ-C30 (The European Organization for Research and Treatment of Cancer quality of life questionnaire) and QLQ-CR29 (European Organisation for Research and Treatment of Cancer questionnaire module for colorectal cancer), and HADS. The EuroQol-5D is a generic HRQoL questionnaire which has demonstrated good psychometric properties and allow for comparison with other populations. It has been translated and validated in Spanish. This instrument consists of two parts: the first is a description of the state of health in five dimensions: mobility, self-care, usual activities, pain / discomfort and anxiety / depression. Each of these dimensions is measured by three answer options that define different levels of severity. The second is a visual analogue scale in which patients rate their health on a scale displayed in the form of a thermometer (20 mm), whose ends are 0 (worst imaginable health state) to 100 (best state imaginable health). The EORTC QLQ-C30 is a questionnaire for evaluating the HRQoL for cancer patients undergoing treatment, which has shown good validity and reliability in its Spanish adaptation (Cronbach's alpha coefficient of 0.7). It is one of the instruments measuring quality of life in cancer patients most commonly used and allow the comparison of the results obtained in patients with colorectal cancer patients with other cancers. It consists of 30 items, 28 of them with four possible answers (in all, a little, a lot, a lot) and two items with seven Alternative (visual analogue scale where one is "very poor" and seven "excellent"). The timeframe should refer to the previous week. The scores on each scale are transformed so that the final values are between 0 and 100. In addition to this overall score, the instrument consists of three scales: Global health status: in which a high score represents a high performance in terms of overall health; Functional -scale: consists of five subscales of operation: physical, role, emotional, cognitive and social; Symptoms scale consisting of a number of symptoms: fatigue, nausea, vomiting, pain, dyspnea, insomnia, decreased appetite, constipation, diarrhea and financial difficulties. A high score on each of these symptoms represents a high level of symptoms or problems in this area. The QLQ-CR29 was then developed after revising the QLQ-CR38, and was demonstrated internationally to have both sufficient validity and reliability to support its use as a supplement to the EORTC QLQ-C30 to assess patient-reported outcomes during treatment for colorectal cancer in clinical trials and other settings. The QLQ-CR29 contains 29 items, and is described in detail elsewhere. Briefly, there are 18 items addressing gastrointestinal symptoms, pain and problems with micturition, and there are separate scales for the participants with or without a stoma and separate items addressing sexual function for men and women. The response categories for each item are the same as those used in the QLQ-C30.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for the study if they were included in the surgical waiting list of one of the participating hospitals with a diagnosis of surgically resectable colon or rectum cancer. Colon or rectum cancer diagnosis was based on anatomopathological diagnosis after a biopsy by colonoscopy. Inclusion criteria were having diagnosed with colon cancer (up to 15 cm above the anal margin) and rectum (between the anal margin and 15 cm above it), where curative and / or palliative surgery for treatment by first time were applied and who sign the informed consent to participate in the study consent.

Exclusion Criteria:

* Exclusion criteria were colon or rectum in situ cancer, unresectable tumor, severe mental or physical conditions which preclude the patient to respond to questionnaires, terminal patients, patients unable to respond to questionnaires from any cause or who do not give their consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study included patients drawn from 22 hospitals belonging to the Spanish National Health Service (SNS), which covers the majority (99.8%) of the population of Spain. All covered residents have free access to their primary care physician and to the ED of the hospitals. All of the hospitals have similar technological and human resources.
  Patients with a diagnosis of colon or rectum cancer attending the surgical services of any of these hospitals to undergo surgery between June 2010 and December 2012 were informed of the goals of the study and invited to voluntarily participate.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Mortality | up to five years

SECONDARY OUTCOMES:
Number of participants with Readmission | up to five years
Number of participants with Reintervention | up to five years
Changes in health-related quality of life (in the questionnaires employed in the study) | up to five years
Number of participants with Complications | up to five years
Number of participants with Cancer recurrence | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Quintana, PhD, Principal Investigator — Hospital Galdakao-Usansolo

REFERENCES:
- [Derived] Orive M, Barrio I, Lazaro S, Gonzalez N, Bare M, de Larrea NF, Redondo M, Cortajarena S, Bilbao A, Aguirre U, Sarasqueta C, Quintana JM; REDISSEC-CARESS/CCR group. Five-year follow-up mortality prognostic index for colorectal patients. Int J Colorectal Dis. 2023 Mar 9;38(1):64. doi: 10.1007/s00384-023-04358-0. PMID 36892600
- [Derived] Orive M, Anton-Ladislao A, Lazaro S, Gonzalez N, Bare M, Fernandez de Larrea N, Redondo M, Bilbao A, Sarasqueta C, Aguirre U, Quintana JM; REDISSEC-CARESS/CCR group. Anxiety, depression, health-related quality of life, and mortality among colorectal patients: 5-year follow-up. Support Care Cancer. 2022 Oct;30(10):7943-7954. doi: 10.1007/s00520-022-07177-1. Epub 2022 Jun 23. PMID 35737143
- [Derived] Quintana JM, Anton-Ladislao A, Lazaro S, Gonzalez N, Bare M, de Larrea NF, Redondo M, Escobar A, Sarasqueta C, Garcia-Gutierrez S, Aguirre U, Briones E, Group FTRCR. Quality Indicators and Outcomes in a Prospective Cohort of Colorectal Cancer Patients. J Gastrointest Cancer. 2023 Mar;54(1):20-26. doi: 10.1007/s12029-021-00779-8. Epub 2021 Dec 10. PMID 34893952
- [Derived] Gonzalez N, Lorono A, Aguirre U, Lazaro S, Bare M, Redondo M, Briones E, Sarasqueta C, Bilbao A, de Larrea NF, Quintana JM; REDISSEC-CARESS/CCR group. Risk scores to predict mortality 2 and 5 years after surgery for colorectal cancer in elderly patients. World J Surg Oncol. 2021 Aug 26;19(1):252. doi: 10.1186/s12957-021-02356-6. PMID 34446044
- [Derived] Quintana JM, Anton-Ladislao A, Lazaro S, Gonzalez N, Bare M, de Larrea NF, Redondo M, Briones E, Escobar A, Sarasqueta C, Garcia-Gutierrez S; REDISSEC CARESS-CCR (Results and Health Services Research in Colorectal Cancer)- group. Predictors of readmission and reoperation in patients with colorectal cancer. Support Care Cancer. 2020 May;28(5):2339-2350. doi: 10.1007/s00520-019-05050-2. Epub 2019 Sep 4. PMID 31485982
- [Derived] Mar J, Anton-Ladislao A, Ibarrondo O, Arrospide A, Lazaro-Aramburu S, Gonzalez N, Bare M, Escobar A, Redondo M, Quintana JM; REDISSEC-CARESS/CCR group. Stage- and age-adjusted cost-effectiveness analysis of laparoscopic surgery in rectal cancer. Surg Endosc. 2020 Mar;34(3):1167-1176. doi: 10.1007/s00464-019-06867-y. Epub 2019 May 28. PMID 31140003
- [Derived] Orive M, Aguirre U, Gonzalez N, Lazaro S, Redondo M, Bare M, Anula R, Briones E, Escobar A, Sarasqueta C, Garcia-Gutierrez S, Quintana JM; REDISSEC-CARESS/CCR group. Risk factors affecting hospital stay among patients undergoing colon cancer surgery: a prospective cohort study. Support Care Cancer. 2019 Nov;27(11):4133-4144. doi: 10.1007/s00520-019-04683-7. Epub 2019 Feb 22. PMID 30793242
- [Derived] Quintana JM, Anton-Ladisla A, Gonzalez N, Lazaro S, Bare M, Fernandez de Larrea N, Redondo M, Briones E, Escobar A, Sarasqueta C, Garcia-Gutierrez S; REDISSEC-CARESS/CCR group. Outcomes of open versus laparoscopic surgery in patients with colon cancer. Eur J Surg Oncol. 2018 Sep;44(9):1344-1353. doi: 10.1016/j.ejso.2018.05.030. Epub 2018 Jun 6. PMID 29921557
- [Derived] Mar J, Anton-Ladislao A, Ibarrondo O, Arrospide A, Lazaro S, Gonzalez N, Bare M, Callejo D, Redondo M, Quintana JM; REDISSEC-CARESS/CCR group. Cost-effectiveness analysis of laparoscopic versus open surgery in colon cancer. Surg Endosc. 2018 Dec;32(12):4912-4922. doi: 10.1007/s00464-018-6250-9. Epub 2018 Jun 4. PMID 29869084
- [Derived] Arostegui I, Gonzalez N, Fernandez-de-Larrea N, Lazaro-Aramburu S, Bare M, Redondo M, Sarasqueta C, Garcia-Gutierrez S, Quintana JM; REDISSEC CARESS-CCR Group. Combining statistical techniques to predict postsurgical risk of 1-year mortality for patients with colon cancer. Clin Epidemiol. 2018 Mar 6;10:235-251. doi: 10.2147/CLEP.S146729. eCollection 2018. PMID 29563837
- [Derived] Bare M, Alcantara MJ, Gil MJ, Collera P, Pont M, Escobar A, Sarasqueta C, Redondo M, Briones E, Dujovne P, Quintana JM; CARESS-CCR Study Group. Validity of the CR-POSSUM model in surgery for colorectal cancer in Spain (CCR-CARESS study) and comparison with other models to predict operative mortality. BMC Health Serv Res. 2018 Jan 29;18(1):49. doi: 10.1186/s12913-018-2839-x. PMID 29378647
- [Derived] Quintana JM, Gonzalez N, Anton-Ladislao A, Redondo M, Bare M, Fernandez de Larrea N, Briones E, Escobar A, Sarasqueta C, Garcia-Gutierrez S, Aguirre U; REDISSEC-CARESS/CCR group. Colorectal cancer health services research study protocol: the CCR-CARESS observational prospective cohort project. BMC Cancer. 2016 Jul 8;16:435. doi: 10.1186/s12885-016-2475-y. PMID 27391216